CLINICAL TRIAL: NCT01472432
Title: Dipeptidyl Peptidase (DPP) IV Inhibition Facilitates Healing of Chronic Foot Ulcers in Patients With Type 2 Diabetes
Brief Title: DPP IV Inhibition Facilitates Healing of Chronic Foot Ulcers in Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Raffaele Marfella, Assistant Professor, University of Campania Luigi Vanvitelli
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IT 345461
Record Dates: First submitted 2011-11-07; First posted 2011-11-16 (Estimated); Results first posted 2015-06-04 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Foot Ulcers
Keywords: type 2 diabetes; healing; foot ulcers; vildagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Foot Ulcer | interventions — Vildagliptin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): In the placebo group, the dose of other concomitant hypoglycemic medication was changed to obtain a similar profile of metabolic parameters. All patients had diabetes and at least one full-thickness wound below the ankle for >3 months. All patients were examined weekly for the first 4 weeks (day 28) then every other week until day 120 or ulcer closure by any means. At each visit, tracings of the wound margins were made for computer planimetry to document changes in wound size, and photographs were taken for a visual record. All patients followed the regular treatment at the multidisciplinary diabetes foot clinic, included treatment of infection, debridement, off-loading, and metabolic control according to high international standards and standard good medical practice.
  Interventions: Drug: Placebo
- Vildagliptin (Experimental): The experimental arm followed the same treatment of placebo group, but received also vildagliptin 50 mg per os b.i.d. for 4 months
  Interventions: Drug: vildagliptin

INTERVENTIONS:
Drug: Placebo — Placebo is added to the standard good medical practice. Plus Metformin and/or Sulfonylurea
  Arms: Placebo
Drug: vildagliptin — 50 mg per os b.i.d. for 4 months of treatment, added to the standard good medical practice.Plus Metformin and/or Sulfonylurea
  Arms: Vildagliptin

SUMMARY:
A randomized versus placebo trial designed to evaluate the clinical and humoral effects of 4 months of vildagliptin on healing of chronic ulcers in type 2 diabetes.

DETAILED DESCRIPTION:
The chronic foot ulcer is a leading cause of hospital admissions for people with diabetes in the developed world and is a major morbidity associated with diabetes, often leading to pain, suffering, and a poor quality of life for patients. Chronic diabetic foot ulcers are estimated to occur in 15% of all patients with diabetes and precede 84% of all diabetes-related lower-leg amputations.The pathophysiology of chronic diabetic ulcers is complex and still incompletely understood, the most important predisposing factors being diabetic neuropathy and vasculopathy. Both micro and macroangiopathy strongly contribute to development and delayed healing of diabetic wounds, through an impaired tissue feeding and response to ischemia. HIF-1α and VEGF, as well as the NO production from iNOS, may contribute to limitation of hypoxic injury by promoting angiogenesis and wound healing. Experimental and pathological studies suggest that suggest that he incretin hormone glucagon-like peptide-1 (GLP-1) may improves VEGF generation, and promote pancreatic islet viability through the up-regulation of HIF1α.

Therefore, aim of this study is to evaluate the effect of the augmentation of GLP-1, by inhibitors of the dipeptidyl peptidase IV (DPP-4), such as vildagliptin, on HIF-1α, VEGF and iNOS in diabetic chronic ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Oral hypoglycemic agents treatment
* Chronic foot ulcers
* Adequate blood circulation (perfusion) was assessed by a dorsum transcutaneous oxygen test >30 -mmHg, anklebrachial index values > 0.7 and < 1.2 with toe pressure > 30 mmHg, or Doppler arterial aveforms that were triphasic or biphasic at the ankle of the affected leg
* Written consensus

Exclusion Criteria:

* Active Charcot disease
* Ulcers resulting from electrical, chemical, or radiation burns
* Collagen vascular disease
* Ulcer malignancy
* Untreated osteomyelitis, or cellulitis
* Ulcer treatment with normothermic or hyperbaric oxygen therapy
* Concomitant medications such as corticosteroids, immunosuppressive medications, or -chemotherapy
* Recombinant or autologous growth factor products
* Skin and dermal substitutes within 30 days of study start
* Use of any enzymatic debridement treatments
* Pregnant or nursing mothers

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2011-05; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele Marfella, MD, PhD, Principal Investigator — Second University Naples
Locations (1):
- Second university of Naples, Naples, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Marfella R, Sasso FC, Rizzo MR, Paolisso P, Barbieri M, Padovano V, Carbonara O, Gualdiero P, Petronella P, Ferraraccio F, Petrella A, Canonico R, Campitiello F, Della Corte A, Paolisso G, Canonico S. Dipeptidyl peptidase 4 inhibition may facilitate healing of chronic foot ulcers in patients with type 2 diabetes. Exp Diabetes Res. 2012;2012:892706. doi: 10.1155/2012/892706. Epub 2012 Nov 1. PMID 23197976

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Completed
Groups:
- Placebo: In the placebo group, the dose of other concomitant hypoglycemic medication was changed to obtain a similar profile of metabolic parameters. Additional antidiabetic therapy, including sulfonylurea, metformin, and insulin, was titrated for optimal glycemic control for 3 months. All patients had diabetes and at least one full-thickness wound below the ankle for >3 months. All patients were examined weekly for the first 4 weeks (day 28) then every other week until day 120 or ulcer closure by any means. At each visit, tracings of the wound margins were made for computer planimetry to document changes in wound size, and photographs were taken for a visual record. All patients followed the regular treatment at the multidisciplinary diabetes foot clinic, included treatment of infection, debridement, off-loading, and metabolic control according to high international standards and standard good medical practice.
  placebo: Placebo is added to the standard good medical practice.
- Vildagliptin: The experimental arm followed the same treatment of placebo group, but received also vildagliptin 50 mg per os b.i.d. for 4 months
  vildagliptin: 50 mg per os b.i.d. for 4 months of treatment, added to the standard good medical practice.
Period: Overall Study
Arm/Group | Placebo | Vildagliptin
Started | 53 | 53
Ulcer Reduction | 13 | 33
Completed | 53 | 53
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Vildagliptin | Total
Number analyzed (Participants) | 53 | 53 | 106
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 12 | 25
  >=65 years | 40 | 41 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] — The study group comprised 106 type 2 diabetic with chronic non-healing diabetic foot ulcers for more than 3 months duration. Patients were enrolled in the study between December 2008 and March 2011. Fifty-three diabetic patients were randomized (simple randomization, open labeled) to receive vildagliptin (50 mg b.i.d., n= 53) in addition to other concomitant hypoglycemic medication for 3 months.
  years | 63 (14) | 64 (15) | 64 (21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 37
  Male | 34 | 35 | 69
Region of Enrollment [Number; unit: participants]
  Italy | 53 | 53 | 106

OUTCOME MEASURES:

1. Primary Outcome: Full Epithelialization of the Wound
Description: Biopsy is performed from the periphery of the ulcer, before and after treatment with vildagliptin, in order to evaluate the above referred outcome.
  Optic microscopy is used to evaluate the epithelialization of the wound.
Time Frame: 3 months of treatment with vildagliptin
Measure: Number; unit: participants
Arm/Group | Placebo | Vildagliptin
Number analyzed (Participants) | 53 | 53
participants | 16 | 8
Statistical Analysis 1: Comparison: Placebo vs Vildagliptin; * Vildagliptin vs Placebo at 3 months. * Placebo baseline versus placebo 3 months. * Vildagliptin baseline versus Vildagliptin 3 months; Test type: Superiority or Other; p < 0.05, t-test, 2 sided — * Vildagliptin vs Placebo at 3 months. * Placebo baseline versus placebo 3 months. * Vildagliptin baseline versus Vildagliptin 3 months; * Vildagliptin vs Placebo at 3 months. * Placebo baseline versus placebo 3 months. * Vildagliptin baseline versus Vildagliptin 3 months

2. Primary Outcome: Capillary Density
Description: Biopsy is performed from the periphery of the ulcer, before and after treatment with vildagliptin, in order to evaluate the above referred outcome.
  Capillary density is measured using immunohistochemistry
Time Frame: 3 months of treatment with vildagliptin
Measure: Median (Inter-Quartile Range); unit: capillaries/mm2
Arm/Group | Placebo | Vildagliptin
Number analyzed (Participants) | 53 | 53
capillaries/mm2
  3 months data | 50 [20 to 90] | 140 [100 to 180]
  baseline data | 48 [15 to 80] | 46 [12 to 88]
Statistical Analysis 1: Comparison: Placebo vs Vildagliptin; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.05, t-test, 2 sided — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: HIF-1α
Description: The factor is assessed by immunoblot analysis (commercial kits). Arbitrary unit of measure are used to evaluate HIF-1α concentration. Higher values represent more factor.
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: arbitrary units
Arm/Group | Placebo | Vildagliptin
Number analyzed (Participants) | 53 | 53
arbitrary units
  3 months data | 200 [150 to 400] | 600 [380 to 800]
  Baseline data | 205 [96 to 350] | 215 [60 to 400]
Statistical Analysis 1: Comparison: Placebo vs Vildagliptin; p-values from multiple comparisons: placebo at baseline vs. placebo at 3 months; placebo at 3 months vs. Vildagliptin at 3 months; Vildagliptin at baseline vs. Vildagliptin at 3 months; Test type: Superiority or Other; p < 0.05, t-test, 2 sided — P-values from multiple comparisons: placebo at baseline vs. placebo at 3 months; placebo at 3 months vs. Vildagliptin at 3 months; Vildagliptin at baseline vs. Vildagliptin at 3 months. P< 0.05 versus control patients. P < 0.05 versus baseline

4. Secondary Outcome: VEGF
Description: The factor is assessed by immunoblot analysis (commercial kits).Arbitrary unit of measure are used to evaluate VEGF concentration. Higher values represent more factor.
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: arbitrary units
Arm/Group | Placebo | Vildagliptin
Number analyzed (Participants) | 53 | 53
arbitrary units
  3 months data | 200 [100 to 500] | 580 [200 to 900]
  Baseline data | 210 [140 to 260] | 215 [160 to 280]
Statistical Analysis 1: Comparison: Placebo vs Vildagliptin; Test type: Superiority or Other; p < 0.05, t-test, 2 sided — P< 0.05 versus control patients. P < 0.05 versus baseline

5. Secondary Outcome: VEGF-R1 (Total and Phosphorylated Form), VEGF-R2 (Total and Phosphorylated Form)
Description: The factor is assessed by immunoblot analysis (commercial kits). Arbitrary unit of measure are used to evaluate VEGF-R1 concentration. Higher values represent more factor.
Time Frame: 3 months
Population: The analysis was not performed because an inadequate amount of biopsy tissue
Arm/Group | Placebo | Vildagliptin
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: iNOS
Description: The factor is assessed by immunoblot analysis (commercial kits). Arbitrary unit of measure are used to evaluate iNOS concentration. Higher values represent more factor.
Time Frame: 3 months
Population: The analysis was not performed because an inadequate amount of biopsy tissue
Arm/Group | Placebo | Vildagliptin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 years
Arm/Group | Placebo | Vildagliptin
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/53
Other Adverse Events (participants affected / at risk) | 0/53 | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No